CLINICAL TRIAL: NCT06206499
Title: Laterally Rotated Flap for Soft Tissue Augmentation Around Maxillary Loaded Osseointegrated Dental Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier Rodriguez Lozano, PhD, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2586/2019
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Implant Tissue Failure; Dental Implant Failed; Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laterally Rotated Flap (Experimental): LRF, Moreno and Caffesse, 2016
  Interventions: Procedure: soft tissue augmentation
- Free gingival graft (Active Comparator): FGG, Sullivan and Atkins, 1968, Langer and Sullivan, 1989
  Interventions: Procedure: soft tissue augmentation

INTERVENTIONS:
Procedure: soft tissue augmentation — Laterally Rotated Flap: A Split-thickness recipient bed on the buccal and mesial aspects of the implant was prepared, resulting in a firm attached bleeding area. The extension of the incisions towards the palate and the distance between them are dependent on the amount of keratinized tissue graft needed for each particular case. Habitually, the keratinized tissue is taken from the adjacent crest; however, if needed to displace more tissue, the incisions may be extended into the palatal tissue. The flap was prepared partial thickness, and released apically from the periosteum to allow passive displacement, and suturing without tension. It was latero-mesially displaced with a 90º rotation. The pedicle was sutured to the recipient bed.
  Control group: The surgical procedure followed the design proposed by Sullivans & Atkins 1968 for soft tissue augmentation around teeth and modified by for application around oseointegrated dental implants.

SUMMARY:
Peri-implant mucositis is one of the most common peri-implant diseases. It was reported in more than 20% of the subjects rehabilitated with dental implants (Lee et al. 2017; Rodrigo et al. 2018; Wada et al. 2019). Furthermore, a significant association was found between peri-implant mucositis, and smoking, implant maintenance and peri-implant soft tissue characteristics (Wada et al. 2019).

Soft tissue quality and volume of the peri-implant mucosa are considered important factors in the prognosis of osseointegrated implants. Linkevicius et al. showed that if its soft tissue thickness was less than 2 mm, crestal bone loss might occur (Linkevicius et al. 2009). In addition, when soft tissue width was evaluated, a wider soft tissue band was related to minimal bone remodeling (Linkevicius et al. 2015). Lin et al. reported in a systematic review and meta-analysis that a lack of keratinized tissue (KT) around osseintegrated implants was associated with plaque accumulation, peri-implant tissue inflammation, soft tissue recession and attachment loss (Lin et al. 2013). Moreover, recent studies established the need of a minimal band of 2 mm of KT around osseointegrated implants, and showed that a band less than 2 mm was associated with more brushing discomfort, plaque accumulation, tissue inflammation and marginal bone apical displacement, concluding that a KT>2 mm had a protective effect on peri-implant tissues (Souza et al. 2015, Perussolo et al. 2018, Monje et al. 2019). Furthermore, peri-implant tissue diseases have also been related to an irregular compliance in situations of lack of KT (Monje et al. 2019).

In the presence of peri-implant horizontal and/or vertical soft tissue deficiencias, soft tissue augmentation has been considered a priority, even prior or instead of bone augmentation (Burkhardt et al. 2008, Zucchelli et al. 2013).

ELIGIBILITY:
Inclusion Criteria:

implant with soft tissue recession Plaque index score less than 30% No relevant systemic disease Smokers (Less than 20 cigars/day)

Exclusion Criteria:

Pregnancy-Lactation Relevant systemic disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-04 (Estimated); Primary Completion 2024-09-29 (Estimated); Study Completion 2024-10-29 (Estimated)

PRIMARY OUTCOMES:
Change in soft tissue 6months after procedure | 1 year
  The amount of soft tissue gained in millimeters will be measured before and after

CONTACTS AND LOCATIONS:
Overall Officials: JOSE ANTONIO MORENO RODRÍGUEZ, DDS, Principal Investigator — UNIVERSIDAD DE MURCAI
Locations (1):
- Universidad de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided